CLINICAL TRIAL: NCT00571909
Title: Evaluation and Treatment of Chronic Pain in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Autosomal Dominant Polycystic Kidney Disease (ADPKD) Pain Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Polycystic Kidney Disease Foundation (Other)
Responsible Party: Principal Investigator, Marie Hogan, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-009690; PDK#14 (Other Grant/Funding Number: Polycystic Kidney Disease Foundation)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Kidney, Polycystic, Autosomal Dominant
Keywords: Polycystic Kidney Disease; Chronic Kidney Pain; Autosomal Dominant Polycystic Kidney; Kidney Cyst; VSPL; video thoracoscopic splanchnicectomy
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- video thoracoscopic splanchnicectomy (VSPL) (Experimental)
  Interventions: Procedure: video thorascopic splanchnicectomy (VSPL)

INTERVENTIONS:
Procedure: video thorascopic splanchnicectomy (VSPL) — VSPL is a minimally invasive technique using 1-2cm incisions through which a camera and surgical tools are placed inside the thoracic cavity and the idea of the procedure is to cut the pain pathway linking the splanchnic ganglion with pain centers in the hypothalamus

SUMMARY:
We will enroll 20 patients to evaluate the effectiveness of a new operation known as videothoracoscopic splanchnicectomy (VSPL) for management of chronic kidney pain. This study is being done to test if this procedure is effective in controlling chronic kidney pain.

DETAILED DESCRIPTION:
Some patients with autosomal dominant polycystic kidney disease (ADPKD) have intractable disabling chronic kidney pain. Among methods used to manage these patients, removal of the nerve supply to the kidney by Videothoracoscopic excision of Splanchnic nerve (videothoracoscopic splanchnicectomy - VSPL) is one of the most promising procedures. Few of these procedures have been performed in ADPKD patients (and in only one patient using the less invasive thoracic approach). We recently performed VSPL on two patients who had chronic pain. Both had initial improvement but have had very short follow up. This study should improve understanding of the molecular mechanisms and mediators of kidney pain and provide the hope of an effective procedure to ADPKD patients with chronic kidney pain.

We are now enrolling patients to study the effectiveness of the VSPL operation, collecting information on pain intensity, quality of life, kidney blood flow, kidney/cyst volume and also to study the involved pain pathways.

Baseline Visit - The patient will also have a complete physical exam and have the kidney's filtration rate measured. Urine and blood tests are performed at each evaluation. You will have an MRI performed of your kidneys. There is no radiation exposure associated with this procedure. You will also be asked to complete Quality of Life (QOL), HALT Pain, and Depression Score questionnaires. These will take approximately 15 minutes to complete and will be repeated at each evaluation.

The VSPL operation will be done within approximately 1 week of your Baseline Visit and is considered part of your clinical care and not part of the research.In this procedure the surgeon approaches the nerves supplying the kidneys through the chest wall, using 3 small incisions. He locates these nerves, then cuts a piece of them and removes it from the chest cavity.You will be released from the hospital when your pain is controlled on oral medications.

1 Month Visit-You will be asked to return to the Mayo Clinic one month after your VSPL procedure for a physical exam and completion of the questionnaires.If unable to return to the Mayo Clinic this evaluation can be done with your local doctor.

3 Month Visit-The 3 Month Visit will be identical to the Baseline visit. You will have a physical exam, blood and urine samples, MRI of your kidneys, Iothalamate Clearance, and the three questionnaires to complete.

6 Months: The questionnaires will be mailed to you for completion.

12 Month Visit-The 12 Month Visit is identical to the 1 Month visit. You will be asked to return to the Mayo Clinic for a physical exam and completion of the questionnaires.

2 Year Visit-The 2 Year Visit will be identical to the Baseline visit. You will have a physical exam, blood and urine samples, MRI of your kidneys, measurement of kidney filtration and complete the three questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of Autosomal Dominant Polycystic Kidney Disease (ADPKD)
* History of debilitating kidney pain for at least 6 month. Other methods of pain management will have been appropriately considered and used when feasible and indicated.
* Patient fit for general anesthesia
* Must be able to travel to Mayo Clinic Rochester for 3 visits
* Must be able to cover the cost of the surgery and post operative care.

Exclusion Criteria:

* Pregnant women (must have a confirmed negative pregnancy test)
* Nursing women
* Creatinine > 3mg/dl, or hemodialysis dependent
* Cancer and other major systemic diseases that could prevent follow-up or data interpretation
* Neurologic or psychologic conditions preventing appropriate informed consent
* Uncontrolled hypertension(SBP > 160; DBP >100)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Improvement in pain control and quality of life | 2 yrs

SECONDARY OUTCOMES:
Changes in urine biomarkers compared to pre-operation values within patients will be compared. Changes in kidney volume, kidney cyst volume, and kidney blood flow before and after the operation will be studied. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie C. Hogan, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States